CLINICAL TRIAL: NCT04192253
Title: Treatment of Locally Advanced VULvar CArcinoma in a Neoadjuvant Setting With Carboplatin and Paclitaxel Chemotherapy (VULCANize)
Acronym: VULCANize
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M19VLC
Record Dates: First submitted 2019-11-11; First posted 2019-12-10 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Locally Advanced, Squamous Cell Carcinoma of the Vulva
MeSH Terms: interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: a prospective, phase ll trial to investigate the response rate of carboplatin and paclitaxel in patients with locally advanced vulvar carcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neo-adjuvant Paclitaxel and Carboplatin (Experimental): Paclitaxel 175 mg/m2 and Carboplatin AUC 5 in a 3 weekly schedule
  Interventions: Drug: Paclitaxel and Carboplatin

INTERVENTIONS:
Drug: Paclitaxel and Carboplatin — Paclitaxel 175 mg/m2 and Carboplatin AUC 5 in a 3 weekly schedule

SUMMARY:
Vulvar cancer is a rare malignancy. Surgery is the treatment of choice, but frequently causes invalidating and chronic postoperative morbidity, especially in patients with high stage disease. Theoretically, downstaging with neoadjuvant chemotherapy could shrink the tumour, making surgical treatment less extensive thereby diminishing the chance for morbidity.

DETAILED DESCRIPTION:
Vulvar cancer is a rare malignancy. Surgery is the treatment of choice, but frequently causes invalidating and chronic postoperative morbidity, especially in patients with high stage disease. Theoretically, downstaging with neoadjuvant chemotherapy could shrink the tumour, making surgical treatment less extensive, thereby diminishing the chance for morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Woman k 18 years
* Signed and written informed consent.
* Histologically confirmed squamous cell vulvar carcinoma
* World Health Organization performance status of 0-2
* Adequate hematological function
* Adequate hepatic function
* Adequate renal function
* Negative pregnancy test for woman of childbearing potential
* measurable disease by physical examination
* TNM stage T2, any N, MO

Exclusion Criteria:

* Vulvar cancer other than squamous cell carcinoma at biopsy
* Previous radiotherapy of the vulva, groins or pelvis
* Patients with metastasis limited to the pelvic lymph nodes, who can be primarily operated with curative intent
* Other diagnosis of malignancy or evidence of other malignancy for 5 years before screening for this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — vulva carcinoma
Enrollment: 51 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
tumour size change by neoadjuvant chemotherapy | 18 weeks
  tumour size change by neoadjuvant chemotherapy measured by RECIST 1.1

SECONDARY OUTCOMES:
avoidance of exenterative or invalidating surgery | 21 weeks
  number of patients were surgery can be reduced after the neo-adjuvant chemotherapy
Chemotherapy related morbidity | 21 weeks
  Chemotherapy related morbidity measured by reported adverse events
overall survival | 5 years after treatment
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Amant, MD, PHD, Principal Investigator — NKI-AvL
Locations (1):
- NKI-AVL, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided